CLINICAL TRIAL: NCT02718521
Title: Chinese People's Liberation Army General Hospital
Brief Title: Adequate Hydration Therapy Combined With Intravenous Infusion of Isosorbide Dinitrate Prevention for CIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qian geng, Associate attending doctor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 16kds2
Record Dates: First submitted 2016-03-19; First posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Cardio-Renal Syndrome
Keywords: contrast-induced nephropathy; hydration therapy combined with intravenous infusion of isosorbide; percutaneous coronary intervention
MeSH Terms: conditions — Cardio-Renal Syndrome | interventions — iodixanol; Isosorbide Dinitrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydration Therapy Combined With Isosorbide Dinitrate (Experimental): Intravenous Infusion of Isosorbide Dinitrate 2mg/h combined with normal saline 1 ml/kg·h 6 hours before angiography and 12 hours after angiography
  Interventions: Procedure: Hydration Combined With Intravenous Infusion of Isosorbide Dinitrate; Drug: Visipaque; Drug: 0.9% sodium chloride ﬂuid administration; Drug: isosorbide dinitrate
- Conventional hydration group (Active Comparator): normal saline 0.5 ml/kg·h 6 hours before angiography and 12 hours after angiography
  Interventions: Procedure: Hydration Combined With Intravenous Infusion of Isosorbide Dinitrate; Drug: Visipaque; Drug: 0.9% sodium chloride ﬂuid administration

INTERVENTIONS:
Procedure: Hydration Combined With Intravenous Infusion of Isosorbide Dinitrate — Before the coronary procedures, investigators used the same 0.9% sodium chloride for hydration conbined with isosorbide dinitrate in all patients 6 hours before angiography and 12 hours after angiography
Drug: Visipaque — All study participants received intra-arterial (320 mg I/ml; GE Healthcare)
Drug: 0.9% sodium chloride ﬂuid administration
Drug: isosorbide dinitrate
  Arms: Hydration Therapy Combined With Isosorbide Dinitrate

SUMMARY:
Patients at moderate and high risk for contrast induced nephropathy (CIN) should receive sufficient hydration before application of contrast to prevent CIN, but hydration could obviously increase the preload for congestive heart failure (CHF) patients. Isosorbide Dinitrate could reduce cardiac preload and afterload by expanding vein and artery.so adequate hydration therapy combined with intravenous infusion of isosorbide dinitrate could better prevent contrast-induced nephropathy theoretically.This prospective, randomized, double-blind, comparative clinical trial randomly selected 264 patients with estimated glomerular filtration rate, (eGFR) <60 ml/min per 1.73 m2 and CHF undergoing coronary angiography to receive either the convention hydration (n=200) or the hydration therapy combined with intravenous infusion of isosorbide dinitrate(n=200).

DETAILED DESCRIPTION:
Investigators enroll 400 patients from February 2016 to February 2017, the principal inclusion criterion included CHF: left ventricular eject fraction (LVEF) <= 50%; moderate to severe chronic kidney disease(CKD) was diagnosed as an eGFR 15 to 59 mL/min per 1.73 m2, calculated via the abbreviated Modification of Diet in Renal Disease (MDRD) study equation from SCr obtained within 72 hours of enrollment, patients were scheduled to undergo diagnostic cardiac angiography or percutaneous coronary interventions. We randomly assigned eligible patients in a 1:1 ratio to either the hydration therapy combined with intravenous infusion of isosorbide dinitrate or a standard hydration administration protocol. hydration therapy combined with intravenous infusion of isosorbide dinitrate refer to give intravenous infusion of isosorbide dinitrate on the basis of fully hydration to reduce cardiac preload.afterload and increase the the tolerance degreen of hydration in chronic heart failure patients. both study groups received intravenous fluids for the same hydration dose. All study participants received intra-arterial Visipaque(320 mg I/ml; GE Healthcare) iso-osmolar contrast medium.

Primary end point of the study was the incidence of CIN: The median peak increase in serum creatinine concentration between day 0 (when contrast was administered) and day 7. Definition of CIN was an absolute increase in serum creatinine (SCr) >0.5 mg/dl or a relative increase >25% compared to baseline SCr. Definition of non-Q-wave myocardial infarction was a creatine kinase-myocardial band enzyme elevation 3 times the upper normal value without new Q waves on the electrocardiogram. Definition of Q-wave myocardial infarction was presence of new pathologic Q waves on an electrocardiogram in conjunction with an elevation in creatine kinase greater than 3 times the normal value. All adverse clinical events as well as study end points were monitored and adjudicated by the independent event committee. Each patient was contacted in every week after administration of the contrast, investigated if dialysis or main cardiovascular events (myocardial infarction,acute heart failure and death), and record any adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. congestive heart failure: objective evidences for decreased left ventricular eject fraction (LVEF) <= 50%;
2. moderate to severe chronic kidney disease was defined as an eGFR 15 to 59 mL/min per 1.73 m2, calculated via the abbreviated Modification of Diet in Renal Disease (MDRD) study equation from SCr obtained within 72 hours of enrollment;
3. patients were scheduled to undergo diagnostic cardiac angiography or percutaneous coronary interventions.

Exclusion Criteria:

1. hemodialysis-dependent patients;
2. complicated with severe short-term progressive disease;
3. Patients < 18 years;
4. pregnancy;
5. emergency cardiac catheterisation (eg, primary percutaneous coronary intervention for ST-segment elevation myocardial infarction);
6. exposure to radiographic contrast media within the previous 7 days;
7. acute decompensated heart failure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Contrast induced nephropathy postoperation | 7 days
  a peak serum creatinine increase of either 0.5 mg/dl or 25% from day 0 through day 7

SECONDARY OUTCOMES:
Composite measure of dialysis or main cardiovascular events | 90 days
  dialysis, myocardial infarction, heart failure and all-cause death

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Chen Y, Hu S, Liu Y, Zhao R, Wang L, Fu G, He Q, Su X, Zheng Y, Qi X, Liu H, Wang J, Gao W, Wang M, Liu S, Zheng X, He B, Yang P, Zhou S, Gao C, Qiu C. Renal tolerability of iopromide and iodixanol in 562 renally impaired patients undergoing cardiac catheterisation: the DIRECT study. EuroIntervention. 2012 Nov 22;8(7):830-8. doi: 10.4244/EIJV8I7A126. PMID 23045301
- [Background] Pannu N, Wiebe N, Tonelli M; Alberta Kidney Disease Network. Prophylaxis strategies for contrast-induced nephropathy. JAMA. 2006 Jun 21;295(23):2765-79. doi: 10.1001/jama.295.23.2765. PMID 16788132
- [Background] Schilp J, de Blok C, Langelaan M, Spreeuwenberg P, Wagner C. Guideline adherence for identification and hydration of high-risk hospital patients for contrast-induced nephropathy. BMC Nephrol. 2014 Jan 6;15:2. doi: 10.1186/1471-2369-15-2. PMID 24393347
- [Background] Mehran R, Aymong ED, Nikolsky E, Lasic Z, Iakovou I, Fahy M, Mintz GS, Lansky AJ, Moses JW, Stone GW, Leon MB, Dangas G. A simple risk score for prediction of contrast-induced nephropathy after percutaneous coronary intervention: development and initial validation. J Am Coll Cardiol. 2004 Oct 6;44(7):1393-9. doi: 10.1016/j.jacc.2004.06.068. PMID 15464318
- [Background] Balemans CE, Reichert LJ, van Schelven BI, van den Brand JA, Wetzels JF. Epidemiology of contrast material-induced nephropathy in the era of hydration. Radiology. 2012 Jun;263(3):706-13. doi: 10.1148/radiol.12111667. Epub 2012 Apr 24. PMID 22535561
- [Background] Qian G, Fu Z, Guo J, Cao F, Chen Y. Prevention of Contrast-Induced Nephropathy by Central Venous Pressure-Guided Fluid Administration in Chronic Kidney Disease and Congestive Heart Failure Patients. JACC Cardiovasc Interv. 2016 Jan 11;9(1):89-96. doi: 10.1016/j.jcin.2015.09.026. Epub 2015 Dec 9. PMID 26685074
- [Derived] Qian G, Liu CF, Guo J, Dong W, Wang J, Chen Y. Prevention of contrast-induced nephropathy by adequate hydration combined with isosorbide dinitrate for patients with renal insufficiency and congestive heart failure. Clin Cardiol. 2019 Jan;42(1):21-25. doi: 10.1002/clc.23023. Epub 2019 Jan 7. PMID 30054906